CLINICAL TRIAL: NCT05025878
Title: Metabolic Tracing of Tumour and T Cells in the Ascites of Ovarian Cancer Patients
Brief Title: 13C-Glucose Tracing of Tumour and T Cells in the Ascites of Ovarian Cancer Patients.
Acronym: iMETABO
Status: Recruiting | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Van Andel Research Institute (Other); University of Victoria (Other)
Responsible Party: Sponsor
Other Study IDs: H18-03615
Record Dates: First submitted 2021-08-04; First posted 2021-08-27 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer; Ascites
MeSH Terms: conditions — Ovarian Neoplasms; Ascites

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- [U-13C]glucose: All participants consented to the study will receive the [U-13C]glucose infusion and collection of ascites for research.
  Interventions: Dietary Supplement: [U-13C]Glucose

INTERVENTIONS:
Dietary Supplement: [U-13C]Glucose — Patients are intravenously infused with 28g of [U-13C]glucose over a 5 hour period. Briefly, [U-13C]glucose will be provided by intravenous line containing 8g of [U-13C]glucose in 60 mL over 10 min. After 10 minutes, 4g of [U-13C]glucose will be administered over an hour. This process will continue until the patient's ascites is drained, or after 5 hours. We will monitor blood glucose levels during infusions using a continuous glucose monitor.

SUMMARY:
The objective of the study is to investigate the metabolism of cells in the ascites tumour microenvironment of ovarian cancer patients. This observational study involves intravenous infusion of [U-13C]glucose into patients during standard paracentesis.

DETAILED DESCRIPTION:
Participants and Location:

This study will recruit up to 10 patients of at least 18 years of age with ascites due to diagnosed ovarian cancer. Eligible study patients will be screened and recruited at BC Cancer - Victoria. Paracentesis procedure and patient consent will occur at the Island Health - Royal Jubilee Hospital.

Study Design:

Participants meeting the inclusion criteria will be fitted with a continuous glucose monitor (FreeStyle Libre) before proceeding to their scheduled appointment for paracentesis. Labeled glucose will be administered via I.V. at dose of 8g of labeled glucose in 60 mL over 10 min. This is followed by 4g of labeled glucose in 30 mL over an hour.

Sample collection and processing:

During [U-13C]glucose infusions, the ascites specimens will kept on ice. Samples will be collected and analyzed by flow cytometry and mass spectrometry for states of metabolism and metabolite profiles respectively. The ascites fluid will be monitored for changes in metabolite levels.

[U-13C]glucose Product Information:

[U-13C]glucose clinical grade will be compound BC Cancer Pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian cancer
* Any stage or grade of disease
* Ascites fluid that requires draining
* Any treatment regimen
* Primary or recurrent ascites
* Understands the concept of the study and give informed consent.

Exclusion Criteria:

* Participants must not have diabetes or abnormal hemoglobin A1C levels.
* The patient's glucose levels must be between 4 - 11.1 mM before administering an infusion. This is to ensure that patients are within normal blood glucose levels, as described by Diabetes Canada.
* Participants cannot receive chemotherapy treatment during the 5 hour duration of the experiment as it may compromise the integrity of the data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 18 with ascites due to diagnosed ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Achieve [U-13C]Glucose enrichment in the ascites of ovarian cancer patients | Duration of ascites paracentesis (samples collected hourly, up to 5 hours)
  Extracellular [U-13C]Glucose label enrichment in the ascites fluid (measured by mass spectrometry).
Compare glucose uptake and metabolic pathways in different cell populations in the ascites. | Duration of ascites paracentesis (samples collected hourly, up to 5 hours)
  Fractional enrichment of intracellular [U-13C]Glucose and 13C labeled metabolites in T cells, myeloid cells and tumour cells (measured by mass spectrometry).

SECONDARY OUTCOMES:
Correlate metabolic profiles with functionality of T cells found in the ascites. | One time - Duration of ascites paracentesis
  Multi-parametric flow cytometry analysis of glucose uptake, mitochondrial function, T cell phenotypes and function.

CONTACTS AND LOCATIONS:
Locations (1):
- Jennifer Rauw, Victoria, British Columbia, Canada